CLINICAL TRIAL: NCT05860647
Title: A Single Arm Study of Resting State Functional Magnetic Resonance Imaging (Rs-fMRI)-Guided Theta Burst Stimulation (TBS) in Primary Progressive Aphasia (PPA)
Brief Title: Transmagnetic Stimulation Pilot in Primary Progressive Aphasia
Acronym: TMS in PPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A23-078
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Primary Progressive Aphasia
Keywords: transmagnetic stimulation; functional MRI guided Theta Burst Stimulation
MeSH Terms: conditions — Aphasia, Primary Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intermittent theta burst stimulation (Experimental): All subjects will receive treatment with intermittent theta burst stimulation (iTBS). There will be a total of 5 treatments over a 2-week period. All subjects will receive iTBS to the right TGd region. TBS treatment will also be provided for two additional sites within the large-scale brain networks (LSBNs) that is found to contain the greatest number of connectivity anomalies. Total participation will be 8-10 weeks.
  Interventions: Device: Intermittent theta burst stimulation

INTERVENTIONS:
Device: Intermittent theta burst stimulation — MagVenture TMS Therapy with theta burst stimulation. Resting motor threshold: 80%; Number of pulses per session: 1200 pulses; Inter-train interval: 8 seconds; Pulse frequency in burst: 50 Hertz
  Other Names: Transmagnetic stimulation; MagVenture

SUMMARY:
Frontotemporal degeneration (FTD) is a non-Alzheimer's dementia that is the 2nd most common cause of dementia in the United States. FTD may present with focal language symptoms that are clinically described as primary progressive aphasia (PPA). There are two types of PPA associated with FTD-semantic variant primary progressive aphasia (SV-PPA) and nonfluent/agrammatic variant primary progressive aphasia (NFV-PPA). Both diseases are progressive neurodegenerative disease processes that compromise dominant hemisphere large scale brain network function, ultimately resulting in mutism. There are currently no FDA-approved treatments for PPA and management is mostly supportive. In combination with resting state functional MRI (rs-fMRI), transcranial magnetic stimulation (TMS) with intermittent theta burst stimulation (iTBS) offers a non-invasive alternative to pharmacotherapy in persons with PPA. In our prior studies of Alzheimer's disease (AD) and Lewy body Dementia (LBD) subjects, investigators have determined that the anterior temporal pole (area TGd and TGv) is an area that is commonly dysfunctional in dementia. The investigators have already embarked upon an fMRI guided study of iTBS in early stage Alzheimer's disease where subjects received a series of 5 treatments to distinct brain regions inclusive of area TGd. The investigators propose a case study of 3 PPA studies where rs-fMRI is applied to the large-scale language networks.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of NFV-PPA and SV-PPA based on criteria (Gorno-Tempini et al., 2011)
2. Prior brain imaging performed
3. Mini Mental Status Exam (MMSE)>10
4. Subjects are between 40-90 years of age

Exclusion Criteria:

1. Non-FTD dementia including, but not limited to Alzheimer's, disease, Lewy body dementia, frontotemporal dementia, vascular dementia, Jakob-Creutzfeldt disease, etc.
2. Inability to tolerate rs-fMRI
3. Contraindication of rs-fMRI due to implants or metal
4. Seizure disorder

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Rosenbloom, MD, Principal Investigator — HealthPartners Neurology; Kashyap Bhavani, PhD,MBBS, Principal Investigator — HealthPartners Neuroscience Research
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intermittent Theta Burst Stimulation
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intermittent Theta Burst Stimulation
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Mini-Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination (MMSE), is a brief cognitive screening tool used to assess cognitive function and detect cognitive impairment. Range: [0-30]. A lower score indicates more cognitive impairment.
  units on a scale | 25.3 (3.21)

OUTCOME MEASURES:

1. Primary Outcome: Connectivity Measures of the Left TGd, 55b, and STV Parcellations at Baseline and Post-treatment
Description: The difference and corresponding 95% confidence interval between follow-up and baseline connectivity measures of the TGd parcellations. Range: -1 to 1.
  Positive values indicate areas where connectivity is higher than healthy controls from the Human Connectome Project.
Time Frame: 6 weeks
Measure: Mean (95% Confidence Interval); unit: correlation
Arm/Group | Intermittent Theta Burst Stimulation
Number analyzed (Participants) | 3
correlation
  L55b | -.06 [-.07 to -.04]
  LTgD | .03 [.02 to .05]
  LSTV | -.01 [-.02 to .01]

2. Post Hoc Outcome: Change in Abnormal Connections of Parcellations
Description: Assessed by calculating the difference and standard deviation between follow-up and baseline of number of abnormal connections of the parcellations. Range: 0-378. There are 378 possible connections of the parcellation. Higher values indicate more abnormal connections of the parcellation pre and post-treatment. The change in the number of abnormal connections of the parcellation is reported.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: abnormal connections
Arm/Group | Intermittent Theta Burst Stimulation
Number analyzed (Participants) | 3
abnormal connections
  L55b | 7 (13.7)
  LTgD | 2 (7)
  LSTV | 3.6 (10.7)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Intermittent Theta Burst Stimulation
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent Theta Burst Stimulation (N=3)
Facial Twitching (Musculoskeletal and connective tissue disorders) | 3 (97)
Headache (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT05860647/Prot_SAP_000.pdf